CLINICAL TRIAL: NCT02731248
Title: Pulse Oximeter Screening for Critical Congenital Heart Disease in Newborns
Brief Title: Pulse Oximeter Screening in Congenital Heart Disease
Acronym: POX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Dilek Dilli, Assoc Prof, Dr. Sami Ulus Children's Hospital
Other Study IDs: SamiUlusCH-CHD
Record Dates: First submitted 2016-04-02; First posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Prospective screening study — Prospective screening study in newborns

SUMMARY:
Pulse oximetry screening of newborn infants increases early detection of critical congenital heart disease and minimises the risk of circulatory collapse before surgery. This study provides an update on the implementation of pulse oximetry screening in Turkey

DETAILED DESCRIPTION:
The early detection of life-threatening, critical congenital heart defects in newborn babies still presents an important clinical challenge. Most defects are amenable to intervention but timely diagnosis (ie, before presentation with cardiovascular collapse or death) is crucial. In high-income countries, examination and, increasingly, antenatal ultrasound have formed the basis of screening, but test accuracy of these procedures is variable and many babies with critical congenital heart defects are discharged before diagnosis. Pulse oximetry screening of newborn infants increases early detection of critical congenital heart disease and minimises the risk of circulatory collapse before surgery. This study provides an update on the implementation of pulse oximetry screening in Turkey

ELIGIBILITY:
Inclusion Criteria:

* Babies within the first 24-72 hours followed up in well baby nurseries
* Babies prior to discharge, if discharged before 24 hours of age,
* Babies ≤5 days and still followed up in well baby nurseries
* Babies born ≥35 gestational weeks

Exclusion Criteria:

* Babies within the first 12 hours of life
* Babies >5 days of life
* Babies with a gestational age of >35 weeks
* Babies with major congenital anomaly except congenial heart disease
* Babies who had a prenatal diagnosis of congenital heart disease

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Babies within the first 24-72 hours followed up in well baby nurseries
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
pulse oximeter positivity | 6 months
  Congenital heart disease detection by pulse oximeter

SECONDARY OUTCOMES:
echocardiographic confirmation | 12 months
  echocardiographic confirmation of congenital heart disease

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Dilli, Assoc Prof, Study Chair — DR sami Ulus Training and Research Hospital
Locations (6):
- Turkey (Türkiye) (6):
  - Dr Sami Ulus Children Hospital, Ankara, Ankara
  - Bursa Sevket Yılmaz Training and Research Hospital, Bursa
  - Ataturk University Medical Faculty, Erzurum
  - Mersin Maternity Hospital, Mersin
  - Mugla Sıtkı Koçman University Medical Faculty, Muğla
  - Urfa Maternity Hospital, Sanliurfa

IPD SHARING:
Plan to Share IPD: No